CLINICAL TRIAL: NCT04354636
Title: Clinical and Radiographic Evaluation After the Use of Silver Modified Atraumatic Restorative Treatment Versus Atraumatic Restorative Treatment in the Management of Occlusal Caries of Primary Molars in Preschool Children: Randomized Clinical Trial
Brief Title: Management of Occlusal Caries Using Silver Modified Atraumatic Restorative Treatment Versus Atraumatic Restorative Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatallah Sameh Ahmed Farouk Abdelhamid, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART_ART
Record Dates: First submitted 2020-04-13; First posted 2020-04-21 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Occlusal Caries
MeSH Terms: interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver modified atraumatic restorative treatment (Experimental): Using silver diamine fluoride incorporated with atraumatic restorative treatment
  Interventions: Drug: Silver modified atraumatic restorative treatment
- Atraumatic restorative treatment (Active Comparator): Using atraumatic restorative treatment without the application of silver diamine fluoride
  Interventions: Other: Atraumatic restorative treatment

INTERVENTIONS:
Drug: Silver modified atraumatic restorative treatment — Silver diamine fluoride that will be applied during atraumatic restorative treatment
  Arms: Silver modified atraumatic restorative treatment
Other: Atraumatic restorative treatment — Using atraumatic restorative treatment without applying silver diamine fluoride
  Arms: Atraumatic restorative treatment

SUMMARY:
Silver modified atraumatic restorative treatment (intervention) or atraumatic restorative treatment (Control) will be used to manage occlusal caries in preschool children then the molars will be evaluated at the interval of 3,6 and 12 months clinically and 6 and 12 months radiographically

DETAILED DESCRIPTION:
Aim of the study:

To evaluate the clinical and radiographic outcomes after the use of silver modified atraumatic restorative treatment versus atraumatic restorative treatment in the management of occlusal caries in primary molars in preschool children.

PICO:

Population:

Preschool children (4-6 years) with occlusal caries in second primary molars.

Intervention:

Silver modified atraumatic restorative treatment

Comparator/Control:

Atraumatic restorative treatment.

Outcomes:

Pain (provoked or spontaneous) OHRQoL(oral health related to quality of life) Parental esthetic perception Failure of restoration Caries density in radiograph

Time:

3, 6 and 12 months

Study design:

A randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* • Patient and parent cooperation and compliance.

  * Children aged 4 - 6 years
  * Second primary molars with occlusal caries.
  * No clinical signs and symptoms of pulp involvement
  * No radiographic abnormalities

Exclusion Criteria:

* • Uncooperative children or parents

  * Children with systemic diseases
  * Children with previous allergies to any of the used materials

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Questioning parent about whether the child have pain between follow up intervals (provoked or spontaneous) | 12 months
  Pain reported-Pain history that occurs after treatment at any point (will be recorded at the follow up intervals) Outcome will be binary (yes/no)

SECONDARY OUTCOMES:
OHRQoL(oral health related to quality of life) | 3 months
  The Early Childhood Oral Health Impact Scale (A-ECOHIS) Score 0-52. There will be 13 questions each question with a score 0-5 where 0 = excellent, 1=very good, 2=good, 3=fair , 4=poor and 5= unknown so the less the score the better is the oral health related to quality of life.
Questioning parents about their aesthetic perception | 3 months
  Parent reported (parent is asked whether he/she is accepting the tooth appearance or not) Outcome will be binary (yes/no)
ART assessment criteria (Codes 00-90) | 12 months
  Failure of restoration according to the code in the ART assessment criteria (Codes 00-90).
  Code 00 or 10 are considered successful, codes 11-40 are classified as failures, and codes 50-90 are assigned in case the tooth was unavailable for evaluation
Caries density in radiograph | 12 months
  Pixel grey value

CONTACTS AND LOCATIONS:
Overall Officials: Sherif B El Tawil, Professor, Study Director — Pediatric Dentistry & Dental Public Health Faculty of Dentistry , Cairo university; Dalia M Moheb, Associate professor, Study Director — Pediatric Dentistry & Dental Public Health Faculty of Dentistry , Cairo university
Locations (1):
- Faculty's pediatric dentiatry clinic, Cairo, Gizq, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vollu AL, Rodrigues GF, Rougemount Teixeira RV, Cruz LR, Dos Santos Massa G, de Lima Moreira JP, Luiz RR, Barja-Fidalgo F, Fonseca-Goncalves A. Efficacy of 30% silver diamine fluoride compared to atraumatic restorative treatment on dentine caries arrestment in primary molars of preschool children: A 12-months parallel randomized controlled clinical trial. J Dent. 2019 Sep;88:103165. doi: 10.1016/j.jdent.2019.07.003. Epub 2019 Jul 4. PMID 31279925
- [Background] Saber AM, El-Housseiny AA, Alamoudi NM. Atraumatic Restorative Treatment and Interim Therapeutic Restoration: A Review of the Literature. Dent J (Basel). 2019 Mar 7;7(1):28. doi: 10.3390/dj7010028. PMID 30866534
- [Background] Oliveira BH, Rajendra A, Veitz-Keenan A, Niederman R. The Effect of Silver Diamine Fluoride in Preventing Caries in the Primary Dentition: A Systematic Review and Meta-Analysis. Caries Res. 2019;53(1):24-32. doi: 10.1159/000488686. Epub 2018 Jun 6. PMID 29874642
- [Background] van Gemert-Schriks MC, van Amerongen WE, ten Cate JM, Aartman IH. Three-year survival of single- and two-surface ART restorations in a high-caries child population. Clin Oral Investig. 2007 Dec;11(4):337-43. doi: 10.1007/s00784-007-0138-8. Epub 2007 Aug 21. PMID 17710452